CLINICAL TRIAL: NCT06837987
Title: An Observation of the Safety and Efficacy of a Modified Transplantation Conditioning and aGVHD Prophylaxis for Severe Aplastic Anemia--a Retrospective, Double-center, Single-arm Clinical Study.
Brief Title: Modified Transplantation Regimen and aGVHD Prophylaxis for Severe Aplastic Anemia in the Setting of Allogeneic HSCT.
Acronym: aGVHD
Status: Completed | Type: Observational
Sponsor: Hematology department of the 920th hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KM-08; 202301AY070001-226 (Other Grant/Funding Number: the Joint and Special Project of Kunming medical university)
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Aplastic Anaemia; Transplantation Conditioning
Keywords: modified transplantation conditioning; aplastic anemia; aGVHD prophylaxis
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Modified transplantation system — Modified transplantation conditioning include: Fludarabine 30mg/m2*6 day, Melphalan 100mg/m2*1 day, cyclophosphamide 50mg/kg*2 day.

SUMMARY:
The investigators retrospectively evaluted the safety and efficacy of the modified transplantation conditioning and aGVHD prophylaxis in severe aplastic anemia in 4 transplantation centers.

DETAILED DESCRIPTION:
Aplastic anemia (AA) is a group of myelo-hemopoietic failure syndromes caused by a variety of etiologies. If not intervened, the average expected survival time is less than half a year.Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is one of the possible cures for this disease. The success rate of treatment for this disease can be further improved under the previous regimen system. The survival rate reported in the literature is 60%-90%. From Jun. 2020 to Dec. 2023, 72 patients in 4 transplantation center received this modified transplantation system, The investigators designed this clinical trial to retrospectively evaluted the safety and efficacy of the modified transplantation conditioning and aGVHD prophylaxis in severe aplastic anemia in the 4 clinical center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed with severe aplastic anemia by NCCN guidelines, and has received HSCT with this transplantation preconditioning and aGVHD prophylaxis regimen;
2. Age 3-65 years old;
3. Weight 10Kg-100Kg;
4. Eastern Cooperative Oncology Group (ECOG) score ≤3;
5. No major organ injury (ECG ejection fraction >45%; bilirubin < 2 times the upper limit of normal value; AST and ALT < 3 times the upper limit of normal value; serum creatinine < 2 times the upper limit of normal value);
6. No severe infection;
7. Subjects voluntarily participated in this clinical trial and signed the informed consent.

Exclusion Criteria:

1. Patients with other hematologic diseases who are not eligible for transplantation or who do not wish to receive transplantation;
2. Patients with an expected survival of less than 1 month;
3. Patients with previous autologous or allogeneic hematopoietic stem cell transplantation;
4. pregnant patients;
5. Patients with severe mental or neurological disorders that would affect the ability to provide informed consent and/or to report or observe adverse events;
6. Other conditions that the investigator determines to be inappropriate for enrollment.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with severe aplastic anemia by NCCN guidelines, and has received HSCT with this transplantation preconditioning and aGVHD prophylaxis regimen;
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Primary graft falure rate | From the day of HSCs transfusion to +100 day after HSCT.
  no apperance or complete loss of donor-derived neutrophils by +28 days
aGVHD incidence | From the day of HSCT transfusion to 100 days after HSCT
  proportion of patients who developed aGVHD within 100 days after HSCT

SECONDARY OUTCOMES:
Poor graft function rate | From the day of HSCs transfusion to 24 months after HSCT
  the presence of at least two cytopenic counts beyond +28 days with a transfusion requirement associated with hypoplastic-aplastic bone marrow
cGVHD incidence | From +100 days after HSCT to the follow-up date
  the proportion of patients who developed chronic GVHD within the observation duration
adverse events | From the first day of preconditioning to +100 days after hematopoietic stem cell Transfusion
  the incidence of adverse events during the transplantation preconditioning periods.
2-year Overall survival rate | 24 months
  proportioin of patients who still be alive within 24 months after HSCT
Disease-free survival | 24 months
  proportion of patients still be alive without GVHD or other diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology，920th Hospital of Joint Logistics Support Force, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided